CLINICAL TRIAL: NCT03829306
Title: "Unraveling KAdcyla (Trastuzumab Emtansine; T-DM1) Resistance In HER2-positive Advanced Breast Cancer (ABC): a Prospective GEICAM Study"
Brief Title: Unraveling KAdcyla Resistance In Human Epidermal Growth Factor Receptor 2(HER2) Positive Advanced Breast Cancer (KATIA)
Acronym: KATIA
Status: Completed | Type: Observational
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Roche Farma, S.A (Industry)
Responsible Party: Sponsor
Other Study IDs: GEICAM/2017-04
Record Dates: First submitted 2019-01-10; First posted 2019-02-04 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Advanced Breast Cancer
Keywords: HER2-positive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Primary tumor and/or the recurrence/metastatic prior to receive Kadcyla. Sequential tumor biopsy after 5 days treatment. Metastatic tumor at disease progression.
  Correlative blood samples will be collected for biomarkers analysis at the following extraction times: Baseline (prior to receive Kadcyla), Cycle 2 (pre-dose), Cycle 4 (pre-dose), every 3 cycles (pre-dose) until disease progression and at the end of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aim is to perform a comprehensive and integrated characterization of mechanisms of primary and acquired resistance to Kadcyla in a prospective cohort of progressive/recurrent HER2-positive breast cancer patients.

DETAILED DESCRIPTION:
This exploratory project is a prospective and multicenter study designed to evaluate the mechanisms of primary and acquired resistance to Kadcyla in a cohort of 50 progressive/recurrent HER2+ BC patients planned to be treated with Kadcyla within the approved indication in Spain.

This study will collect high quality molecular data derived from the analysis of serial biological samples (primary tumor and/or metastatic tissue, plasma, serum and whole blood samples), together with annotated clinical follow up, to reach a better understanding of the biological events that drive breast cancer progression and response/resistance to Kadcyla in ABC patients.

ELIGIBILITY:
Inclusion Criteria:

- Patients are eligible to be included in the study only if they meet all of the following criteria and according to the corresponding Summary of Product Characteristics (SmPC):

1. The patient has signed and dated the informed consent form (ICF) and it has been obtained before conducting any study specific procedure.
2. Female or male patients ≥ 18 years of age on day of signing informed consent.
3. Documented HER2-positive breast cancer based on local laboratory determination (preferably assessed on the most recent tumor biopsy available).
4. Patients with evidence of advanced disease not amenable to resection or radiation therapy with curative intent who are planned to receive Kadcyla within the approved indication in Spain: as a single agent for the treatment of adult patients with HER2-positive, unresectable locally advanced or metastatic breast cancer who previously received trastuzumab and a taxane, separately or in combination. Patients should have either:

   * Received prior therapy for locally advanced or metastatic disease, or
   * Developed disease recurrence during or within six months of completing adjuvant therapy
5. Presence of measurable disease according to RECIST 1.1 for assessment of tumor response.
6. Availability of tumor tissue sample from the primary tumor and/or the recurrence/metastatic site. Effort will be made to obtain a biopsy from a metastatic site in easily accessible tissues.
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.
8. Patient must have a life expectancy ≥16 weeks.
9. Resolution of all acute toxic effects of prior anti-cancer therapy or surgical procedures to NCI-CTCAE v5.0 Grade ≤ 1 (except alopecia or other toxicities not considered a safety risk for the patient at investigator´s discretion).
10. Negative serum pregnancy test result for women of childbearing potential and for women who have experienced menopause onset < 12 months prior to study entry.
11. Willingness and ability to comply with the protocol for the duration of the study including tumor and blood sample collection and undergoing the standard medical practice visits.

Exclusion Criteria:

* Patients will be excluded from the study if they meet any of the following criteria and according to the corresponding Summary of Product Characteristics (SmPC):

  1. Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons), within 3 weeks prior to study entry (or a longer period depending on the defined characteristics of the agents used).
  2. Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. Patients with brain metastases may be eligible for the study only if more than 4 weeks elapsed from treatment completion for these metastases (including radiation and/or surgery) and are clinically stable at the time of study entry.
  3. Major surgical procedure unrelated to breast cancer or significant traumatic injury within 28 days prior to study entry or anticipation of the need for major surgery during the period of Kadcyla administration.
  4. To present contraindications for the treatment with Kadcyla according to the corresponding Summary of Product Characteristics (SmPC).
  5. Known hypersensitivity to Kadcyla, excipients and/or murine proteins.
  6. Pregnancy or breast feeding women.
  7. Persistent toxicities ( NCI-CTCAE v 5.0 grade 2) caused by previous cancer therapy (except alopecia or other toxicities not considered a safety risk for the patient at investigator´s discretion).
  8. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
  9. Known active liver disease, for example, due to hepatitis viruses B (HBV), hepatitis viruses C (HCV), autoimmune hepatic disorders, or sclerosing cholangitis.
  10. History of concurrent or previously treated non-breast malignancies except for appropriately treated 1) non-melanoma skin cancer and/or 2) in situ carcinomas, including cervix and colon. A patient with previous invasive non-breast cancer is eligible provided he/she has been disease free for more than 5 years.
  11. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or Kadcyla administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The target population for inclusion in this study is HER2-positive Advanced Breast Cancer patients who are planned to be treated with Kadcyla whithin the approved indication in Spain.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Genomic alterations on tumor samples with Objective Response (OR) to Kadcyla | Estimated median of 12 months (until disease progression is confirmed)
  Genomic alterations at baseline Formalin-Fixed Paraffin-Embedded (FFPE) tumor samples (primary tumor or metastatic sample) will be analysed by F-One. This test provides information about genomic alterations (base substitutions, insertions/deletions, copy number variations and rearrangements) in 315 cancer-related genes plus introns from 28 genes often rearranged or altered in cancer (https://foundationone.com/docs/FoundationOne).
  OR (complete response plus partial response) will be measured in tumor assessments performed approximately every 3 cycles, based on the investigator assessment according to the standard institutional guidelines using RECIST version 1.1.
Tumor-specific mutation in plasma samples with OR to Kadcyla | Estimated median of 12 months (until disease progression is confirmed)
  Tumor-specific mutation identification will be measured by the test Foundation ACT (F-ACT) on plasma samples collected at baseline and at progression.This test probes 62 cancer-related genes across the 4 classes of genomic alterations (https://www.foundationmedicine.com/genomic-testing/foundation-act). OR (complete response plus partial response) will be measured in tumor assessments performed approximately every 3 cycles, based on the investigator assessment according to the standard institutional guidelines using RECIST version 1.1.

SECONDARY OUTCOMES:
Genomic alterations on tumor samples with progression-free survival (PFS) | Estimated median of 12 months (until disease progression is confirmed)
  Genomic alterations at baseline FFPE tumor samples (primary tumor or metastatic sample) will be analysed by F-One. This test provides information about genomic alterations (base substitutions, insertions/deletions, copy number variations and rearrangements) in 315 cancer-related genes plus introns from 28 genes often rearranged or altered in cancer (http://foundationone.com/docs/FoundationOne).
  Progression-free survival (PFS) to Kadcyla and subsequent treatment lines based on the investigator's assessment at 6 and 12 months.
Tumor-specific mutation in plasma samples with progression-free survival (PFS) | Estimated median of 12 months (until disease progression is confirmed)
  Tumor-specific mutation in plasma samples with OR Tumor-specific mutation identification will be measured by the test Foundation ACT (F-ACT) on plasma samples collected at baseline and at progression.
  Progression-free survival (PFS) to Kadcyla and subsequent treatment lines based on the investigator's assessment
Genomic alterations on tumor samples with Progression-free survival | Estimated median of 12 months (until disease progression is confirmed)
  Genomic alterations at baseline FFPE tumor samples (primary tumor or metastatic sample) will be analysed by F-One. This test provides information about genomic alterations (base substitutions, insertions/deletions, copy number variations and rearrangements) in 315 cancer-related genes plus introns from 28 genes often rearranged or altered in cancer (http://foundationone.com/docs/FoundationOne).
  Progression-free survival (PFS) to Kadcyla and subsequent treatment lines based on the investigator's assessment
Genomic alterations on tumor samples with Time to Progression (TTP) | Estimated median of 12 months (until disease progression is confirmed)
  Genomic alterations at baseline FFPE tumor samples (primary tumor or metastatic sample) will be analysed by F-One. This test provides information about genomic alterations (base substitutions, insertions/deletions, copy number variations and rearrangements) in 315 cancer-related genes plus introns from 28 genes often rearranged or altered in cancer (http://foundationone.com/docs/FoundationOne).
  Time to progression (TTP) to Kadcyla and subsequent treatment lines based on the investigator's assessment.
Tumor-specific mutation in plasma samples with Progression-free survival | Estimated median of 12 months (until disease progression is confirmed)
  Tumor-specific mutation identification will be measured by the test Foundation ACT (F-ACT) on plasma samples collected at baseline and at progression.
  Progression-free survival (PFS) to Kadcyla and subsequent treatment lines based on the investigator's assessment
Tumor-specific mutation in plasma samples Time to Progression (TTP) | Estimated median of 12 months (until disease progression is confirmed)
  Tumor-specific mutation identification will be measured by the test Foundation ACT (F-ACT) on plasma samples collected at baseline and at progression.
  Time to progression (TTP) to Kadcyla and subsequent treatment lines based on the investigator's assessment.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Through study treatment, estimated median of 12 months
  Adverse events will be assessed by standard clinical and laboratory tests (hematology, serum chemistry). Adverse events grade will be defined by the NCI-CTCAE v5.0. Dose/schedule modifications will be also recorded.

OTHER OUTCOMES:
Genomic alterations on tumor samples correlation with overall survival (OS) | Estimated median of 12 months (until disease progression is confirmed)
  Genomic alterations at baseline FFPE tumor samples (primary tumor or metastatic sample) will be analysed by F-One. This test provides information about genomic alterations (base substitutions, insertions/deletions, copy number variations and rearrangements) in 315 cancer-related genes plus introns from 28 genes often rearranged or altered in cancer (http://foundationone.com/docs/FoundationOne).
Tumor-specific mutation in plasma samples with overall survival (OS) | Estimated median of 12 months (until disease progression is confirmed)
  Tumor-specific mutation identification will be measured by the test Foundation ACT (F-ACT) on plasma samples collected at baseline and at progression.
Tumor-specific mutation in plasma samples during Kadcyla treatment with clinical benefit to the subsequent lines of therapy in terms of PFS and TTP. | Estimated median of 12 months (until disease progression is confirmed)
  Tumor-specific mutation identification and clonal evolution in correlative plasma samples: Detection of specific gene mutations found in corresponding tissue samples through targeted sequencing (by Illumina MySeq) will be performed on plasma samples at baseline, during Kadcyla treatment and at end of treatment (EOT)/progression. This will be performed using digital Polymerase Chain Reaction (PCR) on circulating tumor DNA (ctDNA) for clonal dynamics monitoring during Kadcyla treatment.
  Progression-free survival (PFS) to Kadcyla and subsequent treatment lines based on the investigator's assessment Time to progression (TTP) to Kadcyla and subsequent treatment lines based on the investigator's assessment.
Serum levels of T-DM1 conjugate and total trastuzumab | Estimated median of 12 months (until disease progression is confirmed)
  Serum levels of T-DM1 conjugate and total trastuzumab (including both conjugated and unconjugated trastuzumab) will be quantified using a validated enzyme-linked immunosorbent assay.
  samples will obtained on cycles 1, 2 and 3: Pre-dose and 30 mins after end-of-Kadcyla infusion
Plasma DM1 concentrations | Estimated median of 12 months (until disease progression is confirmed)
  Plasma DM1 concentrations will be determined by QPS Netherlands BV (Groningen, Netherlands) using a validated liquid chromatography-tandem mass spectrometry method Plasma DM1 concentrations will be determined by QPS Netherlands BV (Groningen, Netherlands) using a validated liquid chromatography-tandem mass spectrometry method. Plasma samples will obtained on cycles 1, 2 and 3: Pre-dose and 30 mins after end-of-Kadcyla infusion
Correlation of genomic alterations detected by 22 gene Next Generation Sequencing (NGS) and FoundationOne® (F-One) on tumor samples and FoundationACT® (F-ACT) in plasma at baseline. | Estimated median of 12 months (until disease progression is confirmed)
Correlation of HER2 amplification levels in tumor between Fluorescence In-Situ Hybridization (FISH) (local and central) and Copy Number Variation (CNV) provided by F-One. | Estimated median of 12 months (until disease progression is confirmed)

CONTACTS AND LOCATIONS:
Overall Officials: Study director, Study Director — Hospital del Mar, Barcelona, Spain; Study director, Study Director — Fundación Jiménez-Díaz, Madrid, Spain
Locations (10):
- Spain (10):
  - Hospital Universitario Virgen Macarena, Seville, Andalusia
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Clínico Universitario "Virgen de la Arrixaca", El Palmar, Murcia
  - Hospital Universitario Santa Creu i Sant Pau, Barcelona
  - ICO L´Hospitalet, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hopsital Clínico San Carlos, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Clínico Universitario de Valencia, Valencia